# Proefpersoneninformatie voor deelname aan medisch-wetenschappelijk onderzoek

#### Invloed cannabis en oxycodon op de ademhaling

Officiële titel: Invloed van  $\Delta 9$ -tetrahydrocannabinol (THC) op oxycodon-geïnduceerde ademhalingsdepressie in gezonde vrijwilligers

### Inleiding

Geachte heer/mevrouw,

Met deze informatiebrief willen we u vragen of u wilt meedoen aan medisch-wetenschappelijk onderzoek. Meedoen is vrijwillig. U leest hier om wat voor onderzoek het gaat, wat het voor u betekent, en wat de voordelen en nadelen zijn. Het is veel informatie. Wilt u de informatie doorlezen en beslissen of u wilt meedoen? Als u wilt meedoen, kunt u het formulier invullen dat u vindt in bijlage C.

#### Stel uw vragen

U kunt uw beslissing nemen met de informatie die u in deze informatiebrief vindt. Daarnaast raden we u aan om dit te doen:

- Stel vragen aan de onderzoeker die u deze informatie geeft.
- Praat met uw partner, familie of vrienden over dit onderzoek.
- Stel vragen aan de onafhankelijk deskundige, dr. Elise Sarton.
- Lees de informatie op www.rijksoverheid.nl/mensenonderzoek.

#### 1. Algemene informatie

Het Leids Universitair Medisch Centrum (LUMC) heeft dit onderzoek opgezet. Hieronder noemen we het LUMC steeds de 'opdrachtgever'. Onderzoekers, dit kunnen artsen, onderzoekers of verpleegkundigen zijn, voeren het onderzoek uit in het LUMC. Voor dit onderzoek zijn 20 proefpersonen nodig. De medisch-ethische toetsingscommissie Leiden-Den Haag-Delft heeft dit onderzoek goedgekeurd.

#### 2. Wat is het doel van het onderzoek?

In dit onderzoeken bekijken we het effecten van medicinale cannabis (met de actieve stof THC) en oxycodon op de ademhaling. Medicinale cannabis wordt steeds vaker gebruikt bij verschillende aandoeningen, waaronder pijn. Het is belangrijk de balans tussen werking en bijwerking van medicijnen goed te onderzoeken. In dit onderzoek bekijken we de effecten van de pijnstiller oxycodon en medicinale cannabis, omdat de combinatie steeds vaker door patiënten wordt gebruikt.

#### 3. Wat is de achtergrond van het onderzoek?

Sterke pijnstillers zoals oxycodon hebben ook een dempend effect op de ademhaling. Dat betekent dat bij teveel of onjuist gebruik, patiënten een ontregelde ademhaling kunnen krijgen. Deze ongewenste bijwerking kan levensbedreigend zijn. Daarnaast wordt oxycodon steeds vaker gebruikt in combinatie met medicinale cannabis. Medicinale cannabis heeft veel effecten, waaronder pijnstilling. Het is niet bekend of en hoe medicinale cannabis en oxycodon elkaar beïnvloeden op het gebied van pijnstilling en/of effecten op de ademhaling. In dit onderzoek bekijken we daarom wat de effecten van medicinale cannabis en oxycodon op pijnstilling en de ademhaling zijn. We onderzoeken dit bij gezonde vrijwilligers die in het verleden ervaring hebben gehad met het gebruik van recreatieve cannabis.

#### 4. Hoe verloopt het onderzoek?

Hoelang duurt het onderzoek?

Doet u mee met het onderzoek? Dan duurt dat in totaal ongeveer 3 weken. In deze weken is 1 bezoek om te bepalen of u geschikt bent om mee te doen en, als u geschikt bent, 2 hele dagen waarop het onderzoek wordt uitgevoerd.

#### Stap 1: bent u geschikt om mee te doen?

We willen eerst weten of u geschikt bent om mee te doen. Daarom doet de onderzoeker een aantal onderzoeken:

- Lichamelijk onderzoek. De onderzoeker luistert naar uw hart en longen en meet uw bloeddruk en hartslag. We meten uw gewicht en lengte.
- Onderzoek naar uw medische geschiedenis en medicijngebruik

U kunt niet meedoen wanneer u meer dan 21 glazen alcohol per week gebruikt. Ook wanneer u in de 4 weken voorafgaand aan de onderzoeksdagen cannabis heeft gebruikt, kunt u niet meedoen met het onderzoek. Let op: het kan voorkomen dat u gezond bent, maar dat u toch niet geschikt bent om mee te doen. De onderzoeker zal u daar meer over vertellen.

#### Stap 2: onderzoeksdagen

Voor het onderzoek is het nodig dat u 2 keer in 2 weken naar het LUMC komt. De twee onderzoeksdagen zijn steeds bijna hetzelfde, ze verschillen alleen in het geneesmiddel dat u inneemt. Een bezoek duurt een hele dag. U komt nuchter naar onze onderzoekslocatie. Dat wil zeggen dat u in de 6 uur voor het bezoek niets mag eten of drinken.

We doen de volgende onderzoeken:

- Lichamelijk onderzoek. De onderzoeker luistert bijvoorbeeld naar uw hart en longen en meet uw bloeddruk.
- U krijgt een drugstest (hiervoor geeft u wat urine af in een potje) en alcoholtest (via een ademtest). Dit kan op de onderzoekslocatie. Als u recent drugs of alcohol heeft gebruikt, wordt de onderzoeksdag afgebroken.

- Voor vrouwen in de vruchtbare leeftijd: u krijgt een zwangerschapstest. Hiervoor geeft u
  wat urine af in een potje. Dit kan op de onderzoekslocatie. Tijdens dit onderzoek mag u
  niet zwanger zijn.
- U krijgt twee infuuslijnen (slangetjes in een bloedvat) in uw arm: één in een ader en één in een slagader. Uit het infuus in de slagader wordt op een aantal tijdstippen een beetje bloed in een buisje afgenomen. In totaal wordt per bezoek 112 milliliter bloed afgenomen, dit zijn ongeveer 8 eetlepels. Deze hoeveelheid geeft bij volwassenen geen problemen. Ter vergelijking: iemand die bloed geeft bij de bloedbank, geeft per keer 500 milliliter bloed. Met het bloedonderzoek onderzoeken we hoeveel cannabis (THC) of oxycodon u heeft opgenomen.
- U wordt aangesloten op onze apparatuur die uw hartslag, zuurstof en bloeddruk continue zal meten.
- Pijntest. Op een aantal vaste tijdstippen doen we een korte drukpijn test. Deze test zullen we eerst oefenen. Met een staafje wordt op uw hand gedrukt. U geeft aan zodra de druk pijnlijk wordt.
- Ademhalingstest. Op een aantal vaste tijdstippen ademt u een luchtmengsel uit een ballon die een verhoogde hoeveelheid koolzuur bevat (CO<sub>2</sub>). Hierdoor gaat u licht hyperventileren. We meten uw ademhaling vlak nadat u het gasmengsel heeft ingeademd via een kapje over neus en mond.
- Vragenlijsten. Op een aantal vaste tijdstippen vult u vragenlijsten in die gaat over mogelijke bijwerkingen van oxycodon of medicinale cannabis.

U neemt in dit onderzoek drie verschillende geneesmiddelen. U neemt een tablet oxycodon of placebo in met een beetje water. Na 1,5 en na 4,5 uur inhaleert u medicinale cannabis via een verdamper. De placebo is een tablet zonder werkzame stof.

Bij dit onderzoek krijg u de ene onderzoeksdag oxycodon en de andere onderzoeksdag placebo. Loting bepaalt in welke volgorde u oxycodon of placebo krijgt. Om het onderzoek goed uit te voeren, weten u en de onderzoeker niet in welke volgorde u de tabletten krijgt. Als het voor uw gezondheid belangrijk is, kan dit wel worden opgezocht.

Aan het einde van iedere onderzoeksdag verwijderen de infusen en blijft u nog even bij ons om te kijken of u zich goed voelt. Daarna mag u (onder begeleiding) naar huis. Mocht u vanwege medische redenen toch niet naar huis kunnen, is er de mogelijkheid een nacht in het ziekenhuis ter observatie te blijven.

#### 5. Welke afspraken maken we met u?

We willen graag dat het onderzoek goed verloopt. Daarom maken we de volgende afspraken met u:

- U doet tijdens dit onderzoek niet ook nog mee aan een ander medisch-wetenschappelijk onderzoek.
- U gebruikt in de vier weken voorafgaand aan het onderzoek geen cannabis.
- U gebruikt niet meer dan 21 glazen alcohol per week.

- U komt naar iedere afspraak. In de 6 uur voor de onderzoeksdag eet en drinkt u niets.
- U neemt contact op met de onderzoeker in deze situaties:
  - U wilt medicijnen gaan gebruiken. Ook als dit homeopathische middelen zijn, natuurgeneesmiddelen, vitaminen of geneesmiddelen van de drogist.
  - o U wordt in een ziekenhuis opgenomen of behandeld.
  - U krijgt plotseling problemen met uw gezondheid.
  - U wilt niet meer meedoen met het onderzoek.
  - Uw telefoonnummer, adres of e-mailadres verandert.

Vrouwen die zwanger zijn of borstvoeding geven, kunnen niet meedoen aan dit onderzoek.

# 6. Van welke bijwerkingen, nadelige effecten of ongemakken kunt u last krijgen?

Door het onderzoek kunt u last krijgen van de volgende ongemakken of bijwerkingen:

- Door de inname van oxycodon kunt u slaperig worden. Daarnaast neemt de ademhaling af (dit is een belangrijk effect wat we meten), u kunt misselijk worden (te behandelen door een snelwerkend medicijn in uw infuus te geven) en u kunt licht in het hoofd worden.
- Door de inhalatie van medicinale cannabis kunt u ook slaperig worden. Daarnaast kunt u zich 'high' voelen en soms ook misselijk.
- Door de ademhalingstest kunt u kortdurend hoofdpijn krijgen. Dit kunnen we behandelen door paracetamol in uw infuus te geven.
- De pijntest is kortdurend pijnlijk. U geeft zelf aan wanneer de test pijnlijk wordt.
- Het prikken van de infusen kan kortdurend pijnlijk zijn. Bij het verwijderen van de infusen, drukken we de insteekopening goed af, toch kunt u daar een blauwe plek aan overhouden. Deze verdwijnt binnen enkele dagen.

# 7. Wat zijn de voordelen en de nadelen als u meedoet aan het onderzoek?

Meedoen aan het onderzoek kan voordelen en nadelen hebben. Hieronder zetten we ze op een rij. Denk hier goed over na, en praat erover met anderen. U heeft zelf geen voordeel van meedoen aan dit onderzoek. Maar met uw deelname helpt u de onderzoekers om meer inzicht te krijgen in de werking van cannabis en oxycodon op de ademhaling.

Meedoen aan het onderzoek kan deze nadelen hebben:

- U kunt last krijgen van de bijwerkingen of nadelige effecten van de geneesmiddelen, zoals beschreven in paragraaf 6.
- U kunt last hebben van de metingen tijdens het onderzoek. Bijvoorbeeld: bloedafname kan wat pijn doen. Of u kunt daardoor een bloeduitstorting krijgen.
- Meedoen aan het onderzoek kost u extra tijd.
- U moet zich houden aan de afspraken die horen bij het onderzoek.

Wilt u niet meedoen?

U beslist zelf of u meedoet aan het onderzoek.

#### 8. Wanneer stopt het onderzoek?

De onderzoeker laat het u weten als er nieuwe informatie over het onderzoek komt die belangrijk voor u is. De onderzoeker vraagt u daarna of u blijft meedoen.

In deze situaties stopt voor u het onderzoek:

- Alle onderzoeken zijn voorbij.
- Het einde van het hele onderzoek is bereikt.
- U bent zwanger geworden.
- U wilt zelf stoppen met het onderzoek. Dat mag op ieder moment. Meld dit dan meteen bij de onderzoeker. U hoeft er niet bij te vertellen waarom u stopt. De onderzoeker kan voor uw veiligheid nog een of meer controles afspreken.
- De onderzoeker vindt het beter voor u om te stoppen. De onderzoeker kan voor uw veiligheid nog een of meer controles afspreken.
- Een van de volgende instanties besluit dat het onderzoek moet stoppen:
  - o het LUMC,
  - o de overheid, of
  - o de medisch-ethische commissie die het onderzoek beoordeelt.

Wat gebeurt er als u stopt met het onderzoek?

De onderzoekers gebruiken de gegevens en het lichaamsmateriaal (bloed) die tot het moment van stoppen zijn verzameld. Als u wilt, kan verzameld lichaamsmateriaal worden vernietigd. Geef dit door aan de onderzoeker. Het hele onderzoek is afgelopen als alle deelnemers klaar zijn.

#### 9. Wat gebeurt er na het onderzoek?

Krijgt u de resultaten van het onderzoek?

Ongeveer 1 jaar na uw deelname laat de onderzoeker u weten wat de belangrijkste uitkomsten zijn van het onderzoek. De onderzoeker kan u ook vertellen in welke volgorde u de geneesmiddelen heeft gekregen. Wilt u dit niet weten? Zeg dat dan tegen de onderzoeker. Hij zal het u dan niet vertellen.

#### 10. Wat doen we met uw gegevens en lichaamsmateriaal?

Doet u mee met het onderzoek? Dan geeft u ook toestemming om uw en lichaamsmateriaal te verzamelen, gebruiken en bewaren.

Welke gegevens bewaren we?

We bewaren deze gegevens:

- uw naam
- uw geslacht
- uw adres
- gegevens over uw gezondheid
- (medische) gegevens die we tijdens het onderzoek verzamelen

#### Welk lichaamsmateriaal bewaren we?

We bewaren buisjes bloed totdat we de hoeveelheid geneesmiddelen hebben gemeten.

Waarom verzamelen, gebruiken en bewaren we uw gegevens en lichaamsmateriaal?

We verzamelen, gebruiken en bewaren uw gegevens en uw lichaamsmateriaal om de vragen van dit onderzoek te kunnen beantwoorden. En om de resultaten te kunnen publiceren.

#### Hoe beschermen we uw privacy?

Om uw privacy te beschermen geven wij uw gegevens en uw lichaamsmateriaal een code. Op al uw gegevens en lichaamsmateriaal zetten we alleen deze code. De sleutel van de code bewaren we op een beveiligde plek in het ziekenhuis. Als we uw gegevens en lichaamsmateriaal verwerken, gebruiken we steeds alleen die code. Ook in rapporten en publicaties over het onderzoek kan niemand terughalen dat het over u ging.

#### Wie kunnen uw gegevens zien?

Sommige personen kunnen wel uw naam en andere persoonlijke gegevens zonder code inzien. Dit zijn mensen die controleren of de onderzoekers het onderzoek goed en betrouwbaar uitvoeren. Deze personen kunnen bij uw gegevens komen:

- Een controleur die voor de opdrachtgever werkt.
- Nationale toezichthoudende autoriteiten. Bijvoorbeeld de Inspectie Gezondheidszorg en Jeugd.

Deze personen houden uw gegevens geheim. Wij vragen u voor deze inzage toestemming te geven.

#### Hoelang bewaren we uw gegevens en lichaamsmateriaal?

We bewaren uw gegevens 25 jaar in het ziekenhuis. Uw bloed wordt onmiddellijk na gebruik (meten van de hoeveelheid geneesmiddelen in het bloed) vernietigd.

#### Kunt u uw toestemming voor het gebruik van uw gegevens weer intrekken?

U kunt uw toestemming voor het gebruik van uw gegevens op ieder moment intrekken. Dit geldt voor het gebruik in dit onderzoek en voor het gebruik in ander onderzoek. Maar let op: trekt u uw toestemming in, en hebben onderzoekers dan al gegevens verzameld voor een onderzoek? Dan mogen zij deze gegevens nog wel gebruiken. Voor uw lichaamsmateriaal geldt dat de onderzoekers dit vernietigen nadat u uw toestemming intrekt. Maar zijn er dan al metingen gedaan met uw lichaamsmateriaal? Dan mag de onderzoeker de resultaten daarvan blijven gebruiken.

#### Wilt u meer weten over uw privacy?

- Wilt u meer weten over uw rechten bij de verwerking van persoonsgegevens? Kijk dan op www.autoriteitpersoonsgegevens.nl.
  - Heeft u vragen over uw rechten? Of heeft u een klacht over de verwerking van uw persoonsgegevens? Neem dan contact op met degene die verantwoordelijk

is voor de verwerking van uw persoonsgegevens. Voor uw onderzoek is dat: het LUMC. Zie bijlage A voor contactgegevens, en website.

Als u klachten heeft over de verwerking van uw persoonsgegevens, raden we u aan om
deze eerst te bespreken met het onderzoeksteam. Bekijk voor meer informatie over
privacy het privacy statement van het LUMC op de LUMC-website: zie bijlage A U kunt
ook naar de Functionaris Gegevensbescherming van het LUMC gaan. Of u dient een
klacht in bij de Autoriteit Persoonsgegevens.

Waar vindt u meer informatie over het onderzoek?

Op de volgende website(s) vindt u meer informatie over het onderzoek. <a href="www.trialregister.nl">www.trialregister.nl</a> Na het onderzoek kan de website een samenvatting van de resultaten van dit onderzoek tonen. U vindt het onderzoek door te zoeken op 'COXY'.

#### 11. Krijgt u een vergoeding als u meedoet aan het onderzoek?

Voor het meedoen aan dit onderzoek krijgt u een onkostenvergoeding van € 400 (bij voltooiing van het gehele onderzoek. Daarnaast krijgt u een vergoeding van de reiskosten. Stopt u vóórdat het onderzoek is afgelopen? Dan krijgt u een lagere vergoeding (à € 10 per deelgenomen uur).

#### 12. Bent u verzekerd tijdens het onderzoek?

Voor iedereen die meedoet aan dit onderzoek is een verzekering afgesloten. De verzekering betaalt voor schade door het onderzoek. Maar niet voor alle schade. In bijlage B vindt u meer informatie over de verzekering en de uitzonderingen. Daar staat ook aan wie u schade kunt melden.

#### 13. We informeren uw huisarts niet

Wij sturen uw huisarts geen brief om te laten weten dat u meedoet aan het onderzoek.

#### 14. Heeft u vragen?

Vragen over het onderzoek kunt u stellen aan de onderzoeker. Wilt u advies van iemand die er geen belang bij heeft? Ga dan naar dr. Elise Sarton. Zij weet veel over het onderzoek, maar werkt niet mee aan dit onderzoek. Heeft u een klacht? Bespreek dit dan met de onderzoeker. Wilt u dit liever niet? Ga dan naar klachtenfunctionaris of de Autoriteit Persoonsgegevens. In bijlage A staat waar u die kunt vinden.

#### 15. Hoe geeft u toestemming voor het onderzoek?

U kunt eerst rustig nadenken over dit onderzoek. Daarna vertelt u de onderzoeker of u de informatie begrijpt en of u wel of niet wilt meedoen. Wilt u meedoen? Dan vult u het toestemmingsformulier in dat u bij deze informatiebrief vindt. U en de onderzoeker krijgen allebei een getekende versie van deze toestemmingsverklaring.

Dank voor uw tijd.

## 16. Bijlagen bij deze informatie

- A. Contactgegevens
- B. Informatie over de verzekering
- C. Toestemmingsformulier

#### Bijlage A: contactgegevens

#### Onderzoekers:

Prof. Dr. Albert Dahan anesthesioloog 071 - 5262301
Dr. Monique van Velzen onderzoeker 071 - 5263359
Drs. Pieter Simons arts-onderzoeker 071 - 5262301
Drs. Jan van Dam arts-onderzoeker 071 - 5262301

Afdeling Anesthesiologie LUMC, H5-P, Albinusdreef 2, 2333 ZA Leiden pijnonderzoek@lumc.nl

#### Onafhankelijk arts:

Dr. Elise Sarton anesthesioloog 071-5266046

#### Klachten:

Bij klachten kunt u zich wenden tot de klachtenfunctionaris van het LUMC via email: klachtenfunctionaris@lumc.nl U kunt ook telefonisch contact opnemen met het secretariaat van Directoraat Kwaliteit en Patiëntveiligheid ( 071-5264646; tijdens kantooruren). Zij zullen u doorverbinden naar de dienstdoende klachtenfunctionaris.

#### Contactgegevens patiëntenservicebureau

LUMC Patiëntenservicebureau Postbus 9600 2300 RC Leiden

Telefoon: 071-5262989

#### Functionaris voor de Gegevensbescherming:

Wanneer u vragen heeft over de bescherming van uw privacy kunt u contact opnemen de functionarissen gegevensbescherming van het LUMC (FG) via <a href="mailto:privacy@lumc.nl">privacy@lumc.nl</a>

Voor meer informatie over uw rechten: Contactgegevens LUMC Albinusdreef 2 2333 ZA Leiden Centraal telefoonnummer: 071 - 5269111

Voor meer informatie over uw rechten zie de website van het LUMC

https://www.lumc.nl/12367/Deelnemers-wetenschappelijk-onderzoek/

#### Bijlage B: informatie over de verzekering

Het LUMC heeft een verzekering afgesloten voor iedereen die meedoet aan het onderzoek. De verzekering betaalt de schade die u heeft doordat u aan het onderzoek meedeed. Het gaat om schade die u krijgt tijdens het onderzoek, of binnen 4 jaar na het onderzoek. U moet schade binnen 4 jaar melden bij de verzekeraar.

Heeft u schade door het onderzoek? Meld dit dan bij deze verzekeraar:

De verzekeraar van het onderzoek is:

Naam: Centramed

Adres: Maria Montessorilaan 9, 2719 DB Zoetermeer

Telefoonnummer: 070-3017070
E-mail: info@centramed.nl

Polisnummer: 624.530.305

De verzekering betaalt maximaal € 650.000 zijn per persoon en € 5.000.000 voor het hele onderzoek (en € 7.500.000 per jaar voor alle onderzoeken van dezelfde opdrachtgever).

Let op: de verzekering dekt de volgende schade niet:

- Schade door een risico waarover we u informatie hebben gegeven in deze brief. Maar dit geldt niet als het risico groter bleek te zijn dan we van tevoren dachten. Of als het risico heel onwaarschijnlijk was.
- Schade aan uw gezondheid die ook zou zijn ontstaan als u niet aan het onderzoek had meegedaan.
- Schade die ontstaat doordat u aanwijzingen of instructies niet of niet goed opvolgde.
- Schade aan de gezondheid van uw kinderen of kleinkinderen.
- Schade door een behandelmethode die al bestaat. Of door onderzoek naar een behandelmethode die al bestaat.

Deze bepalingen staan in het 'Besluit verplichte verzekering bij medisch-wetenschappelijk onderzoek met mensen 2015'. Dit besluit staat in de Wettenbank van de overheid (https://wetten.overheid.nl).

### Bijlage C: toestemmingsformulier proefpersoon

Behorende bij

#### Invloed cannabis en oxycodon op de ademhaling

- Ik heb de informatiebrief gelezen. Ook kon ik vragen stellen. Mijn vragen zijn goed genoeg beantwoord. Ik had genoeg tijd om te beslissen of ik meedoe.
- Ik weet dat meedoen vrijwillig is. Ook weet ik dat ik op ieder moment kan beslissen om toch niet mee te doen met het onderzoek. Of om ermee te stoppen. Ik hoef dan niet te zeggen waarom ik wil stoppen.
- Ik geef de onderzoekers toestemming om mijn gegevens en lichaamsmateriaal te verzamelen en gebruiken. De onderzoekers doen dit alleen om de onderzoeksvraag van dit onderzoek te beantwoorden.
- Ik weet dat voor de controle van het onderzoek sommige mensen al mijn gegevens kunnen inzien. Die mensen staan in deze informatiebrief. Ik geef deze mensen toestemming om mijn gegevens in te zien voor deze controle.

Ik geef toestemming om mij eventueel na dit onderzoek te vragen of

- Ik weet dat ik niet zwanger mag worden tijdens het onderzoek
- Wilt u in de tabel hieronder ja of nee aankruisen?

ik wil meedoen met een vervolgonderzoek.

| | Ik geef de onderzoekers toestemming om na het onderzoek te late weten welke behandeling ik heb gehad. | n<br> | Ja □ | Nee□ |
|---|---|---|---|---|
| - | lk wil meedoen aan dit onderzoek. | | | |
| | n naam is (proefpersoon): | : | _// | _ |
| k verklaar dat ik deze proefpersoon volledig heb geïnformeerd over het genoemde onderzoek. Wordt er tijdens het onderzoek informatie bekend die die de toestemming van de proefpersoon kan beïnvloeden? Dan laat ik dit op tijd weten aan deze proefpersoon. | | | | |
| | am onderzoeker: | : | /_/_ | |
| <br>Эе | <br>proefpersoon kriigt een volledige informatiebrief mee. samen met een getel | <br>kend | e versie \ | <br>⁄an het |

toestemmingsformulier.

Ja □

Nee□